CLINICAL TRIAL: NCT02014480
Title: A Randomized, Double-Blind, 3-Way, Cross-Over Study to Evaluate Lung Function Response After Treatment With Umeclidinium 62.5 mcg, Vilanterol 25 mcg, and Umeclidinium/Vilanterol 62.5/25 mcg Once-Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Cross-Over Study to Evaluate Lung Function Response After Treatment With Umeclidinium (UMEC) 62.5 Micrograms (mcg), Vilanterol (VI) 25 mcg, and Umeclidinium/Vilanterol (UMEC/VI) 62.5/25 mcg Once-Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116132
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Long-acting beta-agonist; Chronic Obstructive Pulmonary Disease; Umeclidinium; Long-acting muscarinic antagonist; Vilanterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Umeclidinium (Experimental): All subjects will receive UMEC in the dose of 62.5 mcg as inhalation powder in the NDPI once daily in the morning over 14 days in a cross over design.
  Interventions: Device: Umeclidinium 62.5 mcg
- Vilanterol (Experimental): All subjects will receive VI in the dose of 25 mcg as inhalation powder in the NDPI once daily in the morning over 14 days in a cross over design.
  Interventions: Device: Vilanterol 25 mcg
- Umeclidinium/Vilanterol (Experimental): All subjects will receive UMEC/VI in the dose of 62.5/25 mcg as inhalation powder in the NDPI once daily in the morning over 14 days in a cross over design.
  Interventions: Device: Umeclidinium/Vilanterol 62.5/25 mcg

INTERVENTIONS:
Device: Umeclidinium 62.5 mcg — Umeclidinium 62.5 mcg once daily in the morning via NDPI.
  Arms: Umeclidinium
Device: Vilanterol 25 mcg — Vilanterol 25 mcg once daily in the morning via NDPI.
  Arms: Vilanterol
Device: Umeclidinium/Vilanterol 62.5/25 mcg — Umeclidinium/Vilanterol 62.5/25 mcg once daily in the morning via NDPI.
  Arms: Umeclidinium/Vilanterol

SUMMARY:
This is a multicenter, randomized, double-blind, 3-way crossover study to evaluate the lung function response to UMEC 62.5 mcg, VI 25 mcg, and UMEC/VI 62.525 mcg, administered once-daily via a novel dry powder inhaler (NDPI) over 14 days in subjects with COPD.

The study consisted of Run in Phase (5 to 7 days), Treatment Phase (made up of 3 treatment periods of 14 days each separated by 10 to 14 days Washout Period) and Follow-up Phase (7 to 9 days after completion of final visit or premature discontinuation). Eligible subjects will be randomized to a sequence of UMEC 62.5 mcg, VI 25 mcg, and UMEC/VI 62.5/25 mcg such that all subjects will receive each treatment.

Serial spirometry assessments will be conducted on Day 1 and Day 14 and trough spirometry will be conducted on Day 2 and Day 15 of each treatment period. On Day 1 and 14 of each treatment period vital signs will be assessed and adverse event (AE)s will be recorded throughout the total duration of the study (approximately 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Type of Patient: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male or female subjects.
* A female is eligible to enter and participate in the study if she is of: Non-child bearing potential. Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, >45 years, in the absence of hormone replacement therapy. OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the acceptable contraceptive methods used consistently and correctly.
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >= 10 pack-years at Visit 1.
* Severity of Disease: A pre- and post-salbutamol FEV1/forced vital capacity (FVC) ratio of <0.70 and a pre- and post-salbutamol FEV1 of <=70% of predicted normal values at Visit 1 calculated using Nutrition Health and Examination Survey (NHANES) III reference Equations.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject, who, in the opinion of the investigator, has any other significant respiratory condition in addition to COPD, should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Allergic rhinitis is not exclusionary. Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary).
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-Lead ECG: An abnormal and significant electrocardiogram (ECG) finding from the 12-lead ECG conducted at Visit 1, Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The study investigator will determine the medical significance of any ECG abnormalities.
* Medication Prior to Spirometry: Unable to withhold salbutamol for the 4 hour period required prior to spirometry testing at each study visit and at each spirometry test performed at home.
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids (12 weeks), oral or parenteral corticosteroids (6 weeks), antibiotics (for lower respiratory tract infection) (6 weeks), cytochrome P450 3A4 strong inhibitors2 (6 weeks), long-acting beta agonist (LABA)/ inhaled corticosteroid (ICS) combination products if LABA/ICS therapy is discontinued completely (30 days), use of ICS at a dose >1000 mcg/day of fluticasone propionate or equivalent (30 days), initiation or discontinuation of ICS use (30 days), tiotropium (7 days), roflumilast (14 days), theophyllines (48 hours), oral leukotriene inhibitors (zafirlukast, montelukast, zileuton) (48 hours), oral beta-agonists long-acting (48 hours), short-acting (12 hours), inhaled long acting beta2-agonists (LABA, e.g., salmeterol, formoterol, indacaterol) (48 hours), LABA/ICS combination products only if discontinuing LABA therapy and switching to ICS monotherapy (48 hours for the LABA component), inhaled sodium cromoglycate or nedocromil sodium (24 hours), inhaled short acting beta2-agonists (4 hours), inhaled short-acting anticholinergic/short-acting beta2-agonist combination products (4 hours) and any other investigational medication 30 days or within 5 drug half-lives (whichever is longer).
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., salbutamol, ipratropium bromide) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2013-02-01; Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Slovakia (5):
  - GSK Investigational Site, Humenné
  - GSK Investigational Site, Kráľovský Chlmec
  - GSK Investigational Site, Poprad
  - GSK Investigational Site, Šaľa
  - GSK Investigational Site, Vráble
- Ukraine (10):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Sympheropol
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 116132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met the eligibility criteria at Screening (Visit 1) completed a 5- to 7-day Run-in Period prior to being randomized to 1 of 6 treatment sequences. The treatment phase was comprised of three 14-day treatment periods, each separated by a 10- to 14-day washout period.
Groups:
- Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg: Participants received umeclidinium (UMEC) 62.5 micrograms (µg), vilanterol trifenatate (VI) 25 µg, and UMEC/VI 62.5/25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day (QD) for 14 days from a Dry Powder Inhaler (DPI). The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg: Participants received VI 25 µg, UMEC/VI 62.5/25 µg, and UMEC 62.5 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg: Participants received UMEC/VI 62.5/25 µg, UMEC 62.5 µg, and VI 25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg: Participants received UMEC 62.5 µg, UMEC/VI 62.5/25 µg, and VI 25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg: Participants received VI 25 µg, UMEC 62.5 µg, and UMEC/VI 62.5/25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg: Participants received UMEC/VI 62.5/25 µg, VI 25 µg, and UMEC 62.5 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
Period: Treatment Period 1 (14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 35 | 35 | 34 | 34 | 35 | 34 (One participant randomized to Sequence 6 actually received UMEC in Treatment Periods 2 and 3.)
Completed | 35 | 34 | 33 | 32 | 34 | 34
Not Completed | 0 | 1 | 1 | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 1 | 0
Period: Washout Period 1 (10 to 14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 35 | 34 | 33 | 32 | 34 | 34
Completed | 35 | 34 | 32 | 32 | 34 | 34
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 2 (14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 35 | 34 | 32 | 32 | 34 | 34
Completed | 34 | 33 | 30 | 31 | 34 | 34
Not Completed | 1 | 1 | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 1 | 0 | 0
Period: Washout Period 2 (10 to 14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 34 | 33 | 30 | 31 | 34 | 34
Completed | 34 | 33 | 30 | 31 | 34 | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 34 | 33 | 30 | 31 | 34 | 34
Completed | 34 | 32 | 29 | 31 | 34 | 32
Not Completed | 0 | 1 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg: All participants received one of the following three treatments in one of three treatment periods QD from the DPI for 14 days: UMEC 62.5 µg inhalation powder; VI 25 µg inhalation powder; and UMEC/VI 62.5/25 µg inhalation powder. Participants were randomized to receive treatment in one of the six following sequences: (1) UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg; (2) VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg; (3) UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg; (4) UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg; (5) VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg; (6) UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg. The three treatment periods were separated by a washout period of 10 to 14 days.
Arm/Group | UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 169
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European Heritage | 207

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Weighted Mean (WM) 0-6 Hour Forced Expiratory Volume in One Second (FEV1) Obtained Post-dose at Day 14 of Each Treatment Period (TP) by Response Type
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM FEV1 was calculated using 0-6 hour post-dose measurements at Day 14 of each TP, which included pre-dose (trough value for Day 14 [mean of the 23 and 24 hour assessments post Day 13 dosing]) and post-dose 15 minutes (min), 30 min, and 1, 3, and 6 hours. BL is the mean FEV1 values recorded 30 min and 5 min pre-dose on Day 1 of each TP, mean BL is the mean of the BLs for each participant, and period BL is the difference between the BL and the mean BL in each TP for each participant. Change from BL for each TP is the Day 14 value minus the BL value for that TP.
Time Frame: Baseline and Day 14 of each treatment period (up to study day 85)
Population: Intent-to-Treat (ITT) Population: all participants (par.) randomized to treatment who received >=1 dose of randomized study medication in a TP. Only par. available at the specified time points were analyzed. Different par. may have been analyzed for different parameters; the overall number of par, analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- UMEC 62.5 µg: Participants received UMEC 62.5 µg inhalation powder QD from the DPI for 14 days during one of the three treatment periods. Each treatment period was followed by a washout period of 10-14 days.
- VI 25 µg: Participants received VI 25 µg inhalation powder QD from the DPI for 14 days during one of the three treatment periods. Each treatment period was followed by a washout period of 10-14 days.
- UMEC/VI 62.5/25 µg: Participants received UMEC/VI 62.5/25 µg inhalation powder QD from the DPI for 14 days during one of the three treatment periods. Each treatment period was followed by a washout period of 10-14 days.
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 202 | 200 | 202
Liters
  Responder to UMEC, n=79, 78, 81 | 0.155 (0.0184) | 0.156 (0.0185) | 0.263 (0.0179)
  Responder to VI, n=78, 77, 80 | 0.135 (0.0182) | 0.182 (0.0183) | 0.264 (0.0180)
  Responder to Neither, n=80, 79, 80 | 0.014 (0.0179) | 0.035 (0.0180) | 0.092 (0.0179)
Statistical Analysis 1: Comparison: UMEC 62.5 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — Analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of treatment, period, mean Baseline, period Baseline, response type and treatment by response type interaction; Mean Difference (Final Values) = 0.108, 95% CI 2-sided [0.065 to 0.151] — Responders to UMEC=responders to UMEC or to both monotherapies, as defined by a participant with an increase from Baseline of >=12% and 200 milliliters (mL) at >=1 time point over 0-6 hours post-dose in FEV1 on Day 1
Statistical Analysis 2: Comparison: VI 25 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.107, 95% CI 2-sided [0.064 to 0.149] — Responders to UMEC=responders to UMEC or to both monotherapies, as defined by a participant with an increase from Baseline of >=12% and 200 mL at >=1 time point over 0-6 hours post-dose in FEV1 on Day 1
Statistical Analysis 3: Comparison: UMEC 62.5 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.129, 95% CI 2-sided [0.086 to 0.171] — Responders to VI=responders to VI or to both monotherapies, as defined by a participant with an increase from Baseline of >=12% and 200 mL at >=1 time point over 0-6 hours post-dose in FEV1 on Day 1
Statistical Analysis 4: Comparison: VI 25 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [0.040 to 0.125] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 5: Comparison: UMEC 62.5 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [0.036 to 0.120] — Responders to Neither=responders to neither UMEC nor VI, as defined by a participant with at least one FEV1 assessment over 0-6 hours post-dose on Day 1 but no increase from Baseline of >=12% and 200 mL at any assessment(s)
Statistical Analysis 6: Comparison: VI 25 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [0.015 to 0.099] — [estimate comment as in outcome 1, analysis 5]

2. Secondary Outcome: Number of Participants (Par.) Who Were Responsive to UMEC/VI, UMEC or, VI According to FEV1 at Day 1 of Each Treatment Period (TP)
Description: A responder is a par. with an increase from BL of >=12% and 200 milliliters (mL) at >=1 time point over 0-6 hours post-dose (PD) in FEV1 on Day 1. A non-responder (NR) is a par. with >=1 FEV1 assessment over 0-6 hours PD on Day 1 but no increase from BL of >=12% and 200 mL at any assessment(s). Missing: no FEV1 data recorded over 0-6 hours PD on Day 1. Response type is defined based on a par.'s response to each individual monotherapy treatment. A responder to UMEC is a par. who is a responder in the UMEC treatment period (TP) and either a NR or has missing data in the VI TP. A responder to VI is a par. who is a responder in the VI TP and either a NR or has missing data in the UMEC TP. A responder to UMEC and VI is a par. who is a responder in both the UMEC and VI TPs. A responder to neither is a par. who is a NR in both the UMEC and VI TPs. Missing: a par. who has missing data in both the UMEC and VI TPs, or who has missing data in one monotherapy period and is a NR in the other.
Time Frame: Baseline (BL) and 0-6 hours post-dose (15 minutes, 30 minutes, and 1, 3, and 6 hours post-dose) on Day 1 of each treatment period (up to study day 66)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 202 | 200 | 202
participants
  Responder | 81 | 81 | 103
  Non-responder | 121 | 119 | 99

3. Secondary Outcome: Number of Participants With a Larger Change From Baseline in 0-6 Hour Weighted Mean FEV1 at Day 14 of Each Treatment Period With UMEC/VI Compared With UMEC and VI Alone
Description: The number of participants with a larger change from Baseline in weighted mean FEV1 with UMEC/VI compared with UMEC and VI alone was recorded. Participants who improved on UMEC/VI had a larger change from Baseline difference in 0-6 hour weighted mean FEV1 on Day 14 on UMEC/VI compared to UMEC or VI alone. Baseline is the mean FEV1 values recorded 30 min and 5 min pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Change from Baseline for each treatment period is the Day 14 value minus the Baseline value for that treatment period.
Time Frame: Baseline and Day 14 of each treatment period (up to study day 85)
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: participants
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 193 | 192 | 0
participants
  Improved on UMEC/VI | 124 | 130 |
  Not improved on UMEC/VI | 69 | 62 |

4. Secondary Outcome: Change From Baseline in Clinic Visit Pre-dose Trough FEV1 at Day 15 of Each Treatment Period
Description: Trough FEV1 on Treatment Day 15 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after dosing on Day 14. Analysis was performed using an ANCOVA model with covariates of treatment, period, mean Baseline (BL), period BL, response type, and treatment by response type interaction. A participant is a reponder to UMEC if they were a responder to UMEC monotherapy or a responder to both UMEC monotherapy and VI monotherapy. A participant is a responder to VI if they were a responder to VI monotherapy or a responder to both UMEC monotherapy or VI monotherapy. BL is the mean FEV1 recorded 30 min and 5 min pre-dose on Day 1 of each treatment period, mean BL is the mean of the BLs for each participant, and period BL is the difference between BL and the mean BL in each treatment period for each participant. Change from BL for each treatment period is the Day 15 value minus the BL value for that treatment period.
Time Frame: Baseline and Day 15 of each treatment period (up to study day 81)
Population: ITT Population. Only those participants available at the specified time points were analyzed. Different participants may have been analyzed for different parameters; the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 202 | 200 | 202
Liters
  Responder to UMEC, n=79, 78, 80 | 0.105 (0.0196) | 0.086 (0.0197) | 0.170 (0.0191)
  Responder to VI, n=78, 78, 80 | 0.088 (0.0194) | 0.106 (0.0193) | 0.166 (0.0191)
  Responder to Neither, n=80, 79, 79 | 0.016 (0.0190) | 0.004 (0.0191) | 0.062 (0.0191)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study medication to the end of treatment (up to Week 24).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Serious Adverse Events (participants affected / at risk) | 1/202 | 1/200 | 1/202
Other Adverse Events (participants affected / at risk) | 5/202 | 10/200 | 10/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 62.5 µg (N=202) | VI 25 µg (N=200) | UMEC/VI 62.5/25 µg (N=202)
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 62.5 µg (N=202) | VI 25 µg (N=200) | UMEC/VI 62.5/25 µg (N=202)
Headache (Nervous system disorders) | 5 | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.